CLINICAL TRIAL: NCT04546581
Title: An International Multicenter, Adaptive, Randomized Double-Blind, Placebo-Controlled Trial of the Safety, Tolerability and Efficacy of Anti-Coronavirus Hyperimmune Intravenous Immunoglobulin for the Treatment of Adult Hospitalized Patients at Onset of Clinical Progression of COVID-19
Brief Title: Inpatient Treatment of COVID-19 With Anti-Coronavirus Immunoglobulin (ITAC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH); International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INSIGHT 013
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: COVID; COVID-19; SARS-CoV-2; SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — HIV hyperimmune globulin; remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive the investigational product and standard of care (SOC).
  Interventions: Biological: Hyperimmune immunoglobulin to SARS-CoV-2 (hIVIG); Drug: Remdesivir
- Control Group (Placebo Comparator): Participants in this group will receive a placebo and standard of care (SOC).
  Interventions: Other: Placebo; Drug: Remdesivir

INTERVENTIONS:
Biological: Hyperimmune immunoglobulin to SARS-CoV-2 (hIVIG) — Hyperimmune immunoglobulin to SARS-CoV-2 (hIVIG) is derived from the plasma of individuals who recover and develop neutralizing antibodies. Participants will receive a single infusion.
  Arms: Intervention Group
Other: Placebo — Participants will receive a single infusion of the placebo (saline).
  Arms: Control Group
Drug: Remdesivir — Remdesivir will be given to participants in both groups as standard of care (SOC).

SUMMARY:
This protocol will serve as a platform for assessing treatments for adult patients hospitalized for medical management of COVID-19 without related serious end-organ failure. Trials will involve sites around the world strategically chosen to ensure rapid enrollment. This trial will compare hyperimmune intravenous immunoglobulin (hIVIG) with matched placebo, when added to standard of care (SOC), for preventing further disease progression and mortality related to COVID-19. SOC will include remdesivir unless it is contraindicated for an individual patient.

DETAILED DESCRIPTION:
The primary endpoint of this trial in hospitalized patients is an ordinal outcome based on the patient's clinical status on Day 7. It includes 7 mutually exclusive categories capturing the range of organ dysfunction that may be associated with progression of COVID-19, such as respiratory dysfunction and coagulation-related complications. The ordinal endpoint is defined as follows:

7. Death

6. End-organ failure

5. Life-threatening end-organ dysfunction

4. Serious end-organ dysfunction

3. Moderate end-organ dysfunction

2. Limiting symptoms due to COVID-19

1. No limiting symptoms due to COVID-19

Secondary endpoints include time to the 3 least favorable categories, time to the 2 most favorable categories, and the pulmonary only and thrombotic only components of the primary ordinal outcome. Mortality, adverse events (AEs), including infusion reactions, and biological correlates of therapeutic activity are also assessed. Because there is no established endpoint for evaluating the clinical efficacy of treatments for COVID-19, other clinically relevant outcomes, including outcomes used in other COVID-19 treatment trials, will be recorded. Thus, the randomized groups (hIVIG + SOC versus placebo + SOC ) can be compared for multiple outcomes, and results can be compared or combined with other trials.

Participants will be randomized (1:1) to a single infusion of hIVIG + SOC or placebo + SOC on the day of randomization (Day 0). Participants taking remdesivir prior to randomization may be enrolled if eligibility criteria are met. Randomized participants who were not taking remdesivir before randomization will start taking remdesivir immediately following the infusion of hIVIG or placebo unless remdesivir is contraindicated. Participants will be followed for 28 days and, if the trial goes to completion, the primary analysis will be completed after all participants are followed for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection documented by polymerase chain reaction (PCR) or other nucleic acid test (NAT) within 3 days prior to randomization OR documented by NAT more than 3 days prior to randomization AND progressive disease suggestive of ongoing SARS-CoV-2 infection
* Symptomatic COVID-19 disease
* Duration of symptoms attributable to COVID-19 ≤ 12 days
* Requiring inpatient hospital medical care for clinical manifestations of COVID-19 (admission for public health or quarantine only is not included)
* Willingness to abstain from participation in other COVID-19 treatment trials until after study Day 7
* Provision of informed consent by participant or legally authorized representative

Exclusion Criteria:

* Prior receipt of SARS-CoV-2 hIVIG or convalescent plasma from a person who recovered from COVID-19 at any time
* Prior receipt of standard IVIG (not hyperimmune to SARS-CoV-2) within 45 days
* Current or predicted imminent (within 24 hours) requirement for any of the following:

  1. Invasive ventilation
  2. Non-invasive ventilation
  3. Extracorporeal membrane oxygenation
  4. Mechanical circulatory support
  5. Continuous vasopressor therapy
* History of allergy to IVIG or plasma products
* History of selective IgA deficiency with documented presence of anti-IgA antibodies
* Any medical conditions for which receipt of the required volume of intravenous fluid may be dangerous to the patient (includes New York Association Class III or IV stage heart failure)
* Any of the following thrombotic or procoagulant disorders:

  1. Acute coronary syndromes, cerebrovascular syndromes and pulmonary or deep venous thrombosis within 28 days of randomization
  2. History of prothrombin gene mutation 20210, homozygous Factor V Leiden mutations, antithrombin III deficiency, protein C deficiency, protein S deficiency or antiphospholipid syndrome
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Neaton, PhD, Principal Investigator — University of Minnesota; Mark Polizzotto, MD, Study Chair — Kirby Institute
Locations (39):
- United States (18):
  - Penrose Hospital, Colorado Springs, Colorado
  - St. Francis Health Services, Colorado Springs, Colorado
  - St. Anthony Hospital, Lakewood, Colorado
  - Saint Anthony North Health Campus, Westminster, Colorado
  - Washington VA Medical Center, Washington D.C., District of Columbia
  - Redmond Regional Medical Center, Rome, Georgia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Hennepin Healthcare Research Institute/HCMC, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - Hendrick Medical Center, Abilene, Texas
  - CHRISTUS Spohn Shoreline Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - CJW Chippenham Medical Center, Richmond, Virginia
  - Henrico Doctors' Hospital (HCA), Richmond, Virginia
- Denmark (8):
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - CHIP, Department of Infectious Diseases, Section 2100, Copenhagen
  - Herlev-Gentofte Hospital, Hellerup
  - Nordsjællands Hospital, Hillerød, Hillerød
  - Hvidovre University Hospital, Department of Infectious Diseases, Hvidovre
  - Kolding Sygehus, Kolding
  - Odense University Hospital, Odense
- Greece (5):
  - Democritus University of Thrace, Alexandroupoli, Thrace
  - 3rd Dept of Medicine, Medical School, NKUA, Athens
  - 1st Respiratory Medicine Dept, Athens University Medical School, Athens
  - Attikon University General Hospital, Athens
  - Dept. of Critical Care & Pulmonary Medicine, Evangelismos General Hospital, Athens
- Japan (2):
  - NCGM, Tokyo
  - Fujita Health University Hospital, Toyoake
- Institute of Human Virology-Nigeria (IHVN), Abuja, Nigeria
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital del Mar, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A public data set will be made available at the end of the trial
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Jha A, Barker D, Lew J, Manoharan V, van Kessel J, Haupt R, Toth D, Frieman M, Falzarano D, Kodihalli S. Efficacy of COVID-HIGIV in animal models of SARS-CoV-2 infection. Sci Rep. 2022 Oct 10;12(1):16956. doi: 10.1038/s41598-022-21223-2. PMID 36216961
- [Derived] ITAC (INSIGHT 013) Study Group. Hyperimmune immunoglobulin for hospitalised patients with COVID-19 (ITAC): a double-blind, placebo-controlled, phase 3, randomised trial. Lancet. 2022 Feb 5;399(10324):530-540. doi: 10.1016/S0140-6736(22)00101-5. Epub 2022 Jan 28. PMID 35093205
- [Derived] Vandeberg P, Cruz M, Diez JM, Merritt WK, Santos B, Trukawinski S, Wellhouse A, Jose M, Willis T. Production of anti-SARS-CoV-2 hyperimmune globulin from convalescent plasma. Transfusion. 2021 Jun;61(6):1705-1709. doi: 10.1111/trf.16378. Epub 2021 Mar 22. PMID 33715160

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 301 | 292
Completed | 288 | 279
Not Completed | 13 | 13
Not completed — Adverse Event | 9 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 301 | 292 | 593
Age, Continuous [Median (Full Range); unit: years] | 58.4 [43.3 to 73.5] | 59.7 [45.9 to 73.5] | 59.0 [44.5 to 73.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 108 | 257
  Male | 152 | 184 | 336
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 39 | 31 | 70
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 40 | 47 | 87
  White | 174 | 160 | 334
  More than one race | 9 | 13 | 22
  Unknown or Not Reported | 36 | 39 | 75

OUTCOME MEASURES:

1. Primary Outcome: Ordinal Outcome Scale - Day 7
Description: The primary objective is to compare the clinical status of patients in each group on day 7 of follow-up using the primary ordinal outcome with 7 mutually exclusive categories:
  7. Death 6. End-organ failure 5. Life-threatening end-organ dysfunction 4. Serious end-organ dysfunction 3. Moderate end-organ dysfunction 2. Limiting symptoms due to COVID-19
  1. No limiting symptoms due to COVID-19
  Outcome is reported as the percent of participants in each of 7 categories. Primary ordinal outcome based on the patient's clinical status on Day 7. It includes 7 mutually exclusive categories capturing the range of organ dysfunction that may be associated with progression of COVID-19, such as respiratory dysfunction and coagulation-related complications.
  Minimum value = 1, Maximum value = 7 Higher scores mean a worse outcome
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 295 | 284
Participants
  Category 7 - Died | 5 | 5
  Category 6 - End organ failure | 9 | 13
  Category 5 - Life threatening end organ dysfunction | 26 | 26
  Category 4 - Serious end organ dysfunction | 25 | 30
  Category 3 - Moderate end organ dysfunction | 32 | 28
  Category 2 - Limiting symptoms due to COVID-19 | 67 | 61
  Category 1 - No limiting symptoms due to COVID-19 | 129 | 116
  Missing | 2 | 5

2. Primary Outcome: Primary Safety Outcome - Death, SAE or Grade 3 or 4 Events Through Day 7
Description: Number of participants with death, SAE or Grade 3 or 4 event through Day 7
Time Frame: Through Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 295 | 284
Participants | 71 | 70

3. Secondary Outcome: N Reaching 3 Least Favorable Categories
Description: N Reaching 3 least favorable categories of ordinal outcome (Categories 5, 6, 7: life-threatening end organ dysfunction, end organ failure, or death)
Time Frame: All of follow-up (through Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 295 | 284
Participants | 45 | 48

4. Secondary Outcome: N Reaching 2 Most Favorable Categories
Description: N Reaching 2 most favorable categories of ordinal outcome (Categories 1 and 2: not requiring oxygen with or without limiting symptoms due to COVID-19)
Time Frame: All of follow-up (through Day 28)
Population: Those in Category 2 at baseline are excluded from this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 219 | 206
Participants | 178 | 160

5. Secondary Outcome: N Discharged or in Most Favorable Category
Description: N discharged from hospital or reaching most favorable ordinal category (category 1: not requiring oxygen and no limiting symptoms due to COVID-19)
Time Frame: All of follow-up (through Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 295 | 284
Participants | 268 | 252

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 18/301 | 22/292
Serious Adverse Events (participants affected / at risk) | 18/301 | 20/292
Other Adverse Events (participants affected / at risk) | 79/301 | 53/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=301) | Control Group (N=292)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
COVID-19 Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=301) | Control Group (N=292)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 5 (6)
Pyrexia (General disorders) | 10 (10) | 5 (6)
Chills (General disorders) | 10 (10) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (6)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3)
Hypotension (Cardiac disorders) | 3 (3) | 1 (1)
Ageusia (General disorders) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Anosmia (General disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decreased appetite (General disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood glucose increased (Endocrine disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dependence on oxygen therapy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea, exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Lethargy (General disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT04546581/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT04546581/SAP_002.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT04546581/ICF_000.pdf